CLINICAL TRIAL: NCT03309020
Title: PREVAIL VII: Persistence of Ebola Virus in Ocular Tissues and Outcomes of Cataract Surgery in Survivors of Ebola Virus Disease
Brief Title: PREVAIL VII: Cataract Surgery in Ebola Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999917167; 17-EI-N167
Record Dates: First submitted 2017-10-12; First posted 2017-10-13 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2020-08-18

CONDITIONS: Cataract
Keywords: OCT; Cataracts; Visual Acuity
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control with clinical need for cataract surgery
  Interventions: Procedure: Cataract surgery
- EVD Survivors (Experimental): EVD survivors with need for cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Cataract surgery and aqueous humor sampling.

SUMMARY:
Objective: Zaire ebolavirus is a single-stranded RNA virus associated with high morbidity and mortality. The most recent epidemic of Ebola virus disease (EVD) in West Africa resulted in over 11,000 deaths and disabling sequelae among survivors, among which eye complications are highly represented. Chronic intraocular inflammation and viral persistence may result in posterior synechiae and cataract formation, resulting in loss of visual acuity and requiring surgical intervention to resolve. Approximately one out of ten Ebola survivors present with cataract, most of whom will require intraocular surgery during their lifetime, and many of whom require intervention in the near future to regain quality of life. For survivors who are blind from cataract, cataract extraction is necessary to restore visual function, allow reintegration into society and facilitate performance of activities of daily living.

However, surgical parameters among Ebola survivors are unknown, including whether Ebola viral RNA persists in aqueous humor, whether additional anti-inflammatory medication is needed, and the expected degree of improvement in visual function. Moreover, sites of viral persistence are unknown, and it is unclear if lens tissues removed during cataract surgery may harbor virus in Ebola-affected eyes. We propose following EVD survivors and control subjects undergoing cataract surgery to determine visual outcomes among Ebola survivors and explore detection of the presence of virus in lens tissues. The data will inform both future surgical intervention and aid in the understanding of the pathophysiology of Ebola-associated eye disease.

Study Population: Up to 60 Ebola survivors and up to 60 controls will be enrolled. The accrual ceiling is 120 participants.

Design: This is a prospective, natural history study to evaluate the persistence of Ebola viral RNA in the eyes of Ebola survivors and assess the response to cataract surgery in survivors as compared to controls. EVD survivors will first undergo assessment of aqueous humor for the presence of viral RNA. Survivors testing negative for viral RNA and control subjects will undergo clinically indicated cataract surgery. Subjects will be evaluated 1 day, 1 week, 1 month, and 3, 6, 9 and 12 months after surgery for safety and visual outcome assessments, and more often as clinically indicated.

Outcome Measures: The primary outcomes are: 1) the proportion of EVD survivors with evidence of persistence of Ebola viral RNA in ocular tissue and 2) the comparison of amount of intraocular inflammation, as measured by average grade of anterior chamber cell by SUN criteria, between EVD survivors and controls at 1 month and 3 months following cataract surgery. Secondary outcomes include: 1) the proportion of survivors with at least 20/40 best corrected visual acuity (BCVA) after cataract surgery, relative to controls; 2) impact of the covariates age and gender on viral persistence and cataract outcomes; 3) post-operative optical coherence tomography results in EVD survivors.

DETAILED DESCRIPTION:
Objective: Zaire ebolavirus is a single-stranded RNA virus associated with high morbidity and mortality. The most recent epidemic of Ebola virus disease (EVD) in West Africa resulted in over 11,000 deaths and disabling sequelae among survivors, among which eye complications are highly represented. Chronic intraocular inflammation and viral persistence may result in posterior synechiae and cataract formation, resulting in loss of visual acuity and requiring surgical intervention to resolve. Approximately one out of ten Ebola survivors present with cataract, most of whom will require intraocular surgery during their lifetime, and many of whom require intervention in the near future to regain quality of life. For survivors who are blind from cataract, cataract extraction is necessary to restore visual function, allow reintegration into society and facilitate performance of activities of daily living.

However, surgical parameters among Ebola survivors are unknown, including whether Ebola viral RNA persists in aqueous humor, whether additional anti-inflammatory medication is needed, and the expected degree of improvement in visual function. Moreover, sites of viral persistence are unknown, and it is unclear if lens tissues removed during cataract surgery may harbor virus in Ebola-affected eyes. We propose following EVD survivors and control subjects undergoing cataract surgery to determine visual outcomes among Ebola survivors and explore detection of the presence of virus in lens tissues. The data will inform both future surgical intervention and aid in the understanding of the pathophysiology of Ebola-associated eye disease.

Study Population: Up to 60 Ebola survivors and up to 60 controls will be enrolled. The accrual ceiling is 120 participants.

Design: This is a prospective, natural history study to evaluate the persistence of Ebola viral RNA in the eyes of Ebola survivors and assess the response to cataract surgery in survivors as compared to controls. EVD survivors will first undergo assessment of aqueous humor for the presence of viral RNA. Survivors testing negative for viral RNA and control subjects will undergo clinically indicated cataract surgery. Subjects will be evaluated 1 day, 1 week, 1 month, and 3, 6, 9 and 12 months after surgery for safety and visual outcome assessments, and more often as clinically indicated.

Outcome Measures: The primary outcomes are: 1) the proportion of EVD survivors with evidence of persistence of Ebola viral RNA in ocular tissue and 2) the comparison of amount of intraocular inflammation, as measured by average grade of anterior chamber cell by SUN criteria, between EVD survivors and controls at 1 month and 3 months following cataract surgery. Secondary outcomes include: 1) the proportion of survivors with at least 20/40 best corrected visual acuity (BCVA) after cataract surgery, relative to controls; 2) impact the of covariates, age and gender on viral persistence and cataract outcomes; 3) post-operative optical coherence tomography results in EVD survivors.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant must be 14 years of age or older.
2. Participant must be able to understand and sign an informed consent or have a parent/legal guardian do so if they are minor children or a legally authorized representative to provide consent for adults without consent capacity.
3. Participant must be either:

   * an Ebola virus disease (EVD) seropositive survivor or seropositive control OR
   * an EVD seronegative survivor or seronegative control (Serology confirmation is available for PREVAIL participants and will be conducted for non-PREVAIL participants.).
4. Participant must have visually significant cataract(s) consistent with level of visual deficit.
5. Participant must have corrected visual acuity worse than 20/40 in affected eye and vision loss believed to be primarily the result of the cataract.
6. Any woman and persons of childbearing potential age have a negative pregnancy test at screening and must be willing to undergo pregnancy testing prior to the cataract surgery.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Concurrent life-threatening illness or other condition that compromises a participant's ability to safely undergo surgery, as determined by the surgical and medical team, including any condition that prevents the participant from lying down supine or remaining still, such as severe lung disease, or a known life-threatening, untreated or unstable cardiac or pulmonary condition.
2. Active uveitis at time of surgery or within the past three months, if documented.
3. Participant is pregnant, as surgery is elective and no adequate data regarding the use of postoperative topical antibiotic-steroid combination drops exists in pregnant women.
4. Any condition that poses a risk to the participant having a safe surgical or post-operative experience, including known inability or unwillingness to follow up for the full duration of the protocol.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M Magone de Quadros Costa, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- PREVAIL JFK Hospital, Monrovia, Liberia

REFERENCES:
- [Result] Eghrari AO, Shantha JG, Ross RD, Ryn CV, Crozier I, Hayek B, Gradin D, Roberts B, Prakalapakorn SG, Amegashie F, Nishant K, Singh G, Dolo R, Fankhauser J, Burkholder B, Pettitt J, Gross R, Brady T, Dighero-Kemp B, Reilly C, Hensley L, Higgs E, Yeh S, Bishop RJ. Efficacy and Safety Outcomes of Cataract Surgery in Survivors of Ebola Virus Disease: 12-Month Results From the PREVAIL VII Study. Transl Vis Sci Technol. 2021 Jan 25;10(1):32. doi: 10.1167/tvst.10.1.32. eCollection 2021 Jan. PMID 33520427

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | EVD Survivors
Started | 12 | 25
Underwent Cataract Surgery | 10 | 24
Completed | 9 | 24
Not Completed | 3 | 1
Not completed — Death | 1 | 0
Not completed — Did not undergo surgery | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | EVD Survivors | Total
Number analyzed (Participants) | 12 | 25 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [40 to 63.8] | 62 [40 to 68] | 59 [40 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 14 | 20
  Male | 6 | 11 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Liberia | 12 | 25 | 37

OUTCOME MEASURES:

1. Primary Outcome: Proportion of EVD Survivors With Evidence of Persistence of Ebola Viral RNA in Ocular Tissue
Description: Participants undergo aqueous fluid (aqueous humor) sampling to assess for the presence of Ebola virus RNA via RT-PCR using the GeneXpert assay.
  The study was intended to include analysis of lens tissue to explore detection of the presence of virus in lens tissue in EVD survivors; however, the collected lens tissue samples were damaged during storage and transport. Therefore, the lens samples were unable to yield any reportable data.
Time Frame: One week prior to cataract surgery
Population: Ebola survivors in the analytic population (seropositive EVD survivors who underwent cataract surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | EVD Survivors
Number analyzed (Participants) | 22
Participants | 0

2. Primary Outcome: Comparison of the Amount of Intraocular Inflammation Between EVD Survivors and Controls at 1 Month Following Cataract Surgery
Description: The amount of intraocular inflammation is measured by the average grade of anterior chamber (AC) cell per Standardization of Uveitis Nomenclature (SUN) criteria.
  AC cell grading, with higher grades indicating a worse outcome:
  Grade 0 -- 0-5 cells per 1 mm x 1 mm high-powered field; Grade 1 -- 6-15 cells per 1 mm x 1 mm high-powered field; Grade 2 -- 16-25 cells per 1 mm x 1 mm high-powered field; Grade 3 -- 26-50 cells per 1 mm x 1 mm high-powered field; Grade 4 -- > 50 cells per 1 mm x 1 mm high-powered field
Time Frame: 1 month after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Mean (Standard Deviation); unit: AC cell grade
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 22
Number analyzed (eyes) | 12 | 22
AC cell grade | .67 (.49) | .64 (.66)
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Null hypothesis is no difference in grade between survivor statuses one month after cataract surgery; Test type: Other; p = 0.802, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment and gender (male or female) were included as covariates in the model

3. Primary Outcome: Comparison of the Amount of Intraocular Inflammation Between EVD Survivors and Controls at 3 Months Following Cataract Surgery
Description: The amount of intraocular inflammation is measured by the average grade of anterior chamber cell per Standardization of Uveitis Nomenclature (SUN) criteria.
  AC cell grading, with higher grades indicating a worse outcome:
  Grade 0 -- 0-5 cells per 1 mm x 1 mm high-powered field; Grade 1 -- 6-15 cells per 1 mm x 1 mm high-powered field; Grade 2 -- 16-25 cells per 1 mm x 1 mm high-powered field; Grade 3 -- 26-50 cells per 1 mm x 1 mm high-powered field; Grade 4 -- > 50 cells per 1 mm x 1 mm high-powered field
Time Frame: 3 months after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Mean (Standard Deviation); unit: AC cell grade
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 22
Number analyzed (eyes) | 12 | 22
AC cell grade | .5 (1.17) | .82 (1.01)
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Null hypothesis is no difference in grade between survivor statuses three months after cataract surgery; Test type: Other; p = .713, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment and gender (male or female) were included as covariates in the model

4. Secondary Outcome: Comparison of Proportion of Eyes With at Least 20/40 Best Corrected Visual Acuity (BCVA) 12 Months After Cataract Surgery
Description: Comparison of proportion with at least 20/40 best corrected visual acuity (BCVA) after cataract surgery 12 months in survivors vs controls. Best corrected visual acuity was measured using the Tumbling-E Early Treatment Diabetic Retinopathy Study (ETDRS) protocol vision chart. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 21
Number analyzed (eyes) | 12 | 21
eyes | 5 | 18
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Null hypothesis is no difference in the proportion of participants with at least 20/40 best corrected visual acuity (BCVA) between survivor statuses; Test type: Other; Odds Ratio (OR) = 0.1, 95% CI 2-sided [0.01 to 0.69] — Odds of eye with at least 20/40 best corrected visual acuity (BCVA) 12 months after cataract surgery for controls vs. EVD survivors

5. Secondary Outcome: Comparison of Intraretinal Fluid Cysts Between EVD Survivors and Controls From Baseline to 12 Months After Cataract Surgery
Description: Optical coherence tomography (OCT) imaging of the retina and optic nerve was used to identify the presence of intraretinal fluid cysts in EVD survivors vs. controls from baseline to 12 months after surgery
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 22
Number analyzed (eyes) | 12 | 22
eyes
  Baseline | 0 | 0
  Month 1 | 0 | 0
  Month 3 | 1 | 3
  Month 6 | 0 | 1
  Month 9 | 1 | 2
  Month 12 | 2 | 2
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Test type: Other; p = .832, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment and gender (male or female) were included as covariates in the model

6. Secondary Outcome: Comparison of Central Subfield Thickness (CST) Between EVD Survivors and Controls From Baseline to 12 Months After Cataract Surgery
Description: Optical coherence tomography (OCT) imaging of the retina and optic nerve was used to measure macular central subfield thickness (CST) in µm in EVD survivors vs. controls from baseline to 12 months after cataract surgery
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: µm
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 22
Number analyzed (eyes) | 12 | 22
µm
  Baseline | 203 [182 to 204] | 209 [184 to 244.5]
  Month 1 | 222 [217.5 to 260] | 224 [211 to 269.5]
  Month 3 | 227 [196.8 to 260.2] | 216 [188 to 253]
  Month 6 | 226.5 [209.5 to 234.8] | 234 [203 to 258]
  Month 9 | 240 [227.8 to 258.2] | 238 [214 to 254.5]
  Month 12 | 244 [221.5 to 264.5] | 231 [212.5 to 245.5]
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Test type: Other; p = .995, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment and gender (male or female) were included as covariates in the model

7. Secondary Outcome: Comparison of Central Subfield Thickness (CST) Between EVD Survivors and Controls, Excluding Cases of Intraretinal Fluid Cysts, From Baseline to 12 Months After Cataract Surgery
Description: Optical coherence tomography (OCT) imaging of the retina and optic nerve was used to measure central subfield thickness (CST) in µm in EVD survivors vs. controls, excluding cases of intraretinal fluid cysts, from baseline to 12 months after cataract surgery
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: µm
Units Other Than Participants: eyes
Arm/Group | Control | EVD Survivors
Number analyzed (Participants) | 8 | 22
Number analyzed (eyes) | 12 | 22
µm
  Baseline | 203 [182 to 204] | 218 [190.2 to 244]
  Month 1 | 222 [217.5 to 260] | 224 [211 to 269.5]
  Month 3 | 223 [196.5 to 248] | 214 [183.5 to 224]
  Month 6 | 220 [207 to 234] | 229 [202.8 to 251.2]
  Month 9 | 240 [225.5 to 253] | 238 [211 to 254]
  Month 12 | 242 [211 to 248] | 231 [216 to 244]
Statistical Analysis 1: Comparison: Control vs EVD Survivors; Test type: Other; p = 0.441, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment and gender (male or female) were included as covariates in the model

8. Secondary Outcome: Impact of Gender on Visual Acuity From Baseline to 12 Months After Surgery
Description: Visual acuity (20/x) was measured using the Tumbling-E Early Treatment Diabetic Retinopathy Study (ETDRS) protocol vision chart. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: visual acuity (20/x)
Units Other Than Participants: eyes
Groups:
- All Participants: EVD Survivors and Control Participants
Arm/Group | All Participants
Number analyzed (Participants) | 30
Number analyzed (eyes) | 34
visual acuity (20/x)
  Baseline | 800 [100 to 4000]
  Month 1 | 40 [25 to 50]
  Month 12 | 32 [25 to 50]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = .892, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Age at enrollment, survivor status (EVD survivor/control) included as covariates; within-subject measurement of distinct eyes treated as independent

9. Secondary Outcome: Impact of Gender on Improvement in the Number of Lines Read on an ETDRS Eye Chart From Baseline to 12 Months After Surgery
Description: Visual acuity was measured using the Tumbling-E Early Treatment Diabetic Retinopathy Study (ETDRS) protocol vision chart. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. Number of lines improvement equals the number of lines read at 12 months post cataract surgery minus the number of lines read at baseline
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: lines of improvement
Units Other Than Participants: eyes
Arm/Group | All Participants
Number analyzed (Participants) | 30
Number analyzed (eyes) | 34
lines of improvement | 8.06 [4.01 to 20.97]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = .913, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 8, analysis 1]

10. Secondary Outcome: Impact of Age on Visual Acuity From Baseline to 12 Months After Surgery
Description: Age was age at enrollment in years. Visual acuity (20/x) was measured using the Tumbling-E Early Treatment Diabetic Retinopathy Study (ETDRS) protocol vision chart. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: visual acuity (20/x)
Units Other Than Participants: eyes
Arm/Group | All Participants
Number analyzed (Participants) | 30
Number analyzed (eyes) | 34
visual acuity (20/x)
  Baseline | 800 [100 to 4000]
  Month 1 | 40 [25 to 50]
  Month 12 | 32 [25 to 50]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = .106, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Gender (male/female), survivor status (EVD survivor/control) as covariates; within-subject measurement of distinct eyes treated as independent

11. Secondary Outcome: Impact of Age on Improvement in the Number of Lines Read on an ETDRS Eye Chart From Baseline to 12 Months After Surgery
Description: Age was age at enrollment in years. Visual acuity was measured using the Tumbling-E Early Treatment Diabetic Retinopathy Study (ETDRS) protocol vision chart. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. Number of lines improvement equals the number of lines read at 12 months post cataract surgery minus the number of lines read at baseline
Time Frame: Baseline to 12 months (1 year) after cataract surgery
Population: Analytic population (seropositive EVD survivors and seronegative controls who underwent cataract surgery)
Measure: Median (Inter-Quartile Range); unit: lines of improvement
Units Other Than Participants: eyes
Arm/Group | All Participants
Number analyzed (Participants) | 30
Number analyzed (eyes) | 34
lines of improvement | 8.06 [4.01 to 20.97]
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.09, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Impact of Gender on Viral Persistence One Week Prior to Cataract Surgery
Description: Participants undergo aqueous fluid (aqueous humor) sampling to assess for the presence of Ebola virus RNA via RT-PCR using the GeneXpert assay.
Time Frame: One week prior to cataract surgery
Population: Zero participants were analyzed due to lack of variability in the outcome (no samples tested positive for viral persistence)
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Impact of Age on Viral Persistence One Week Prior to Cataract Surgery
Description: Age was age at enrollment in years. Participants undergo aqueous fluid (aqueous humor) sampling to assess for the presence of Ebola virus RNA via RT-PCR using the GeneXpert assay.
Time Frame: One week prior to cataract surgery
Population: as for outcome 12
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants are monitored during all study visits, with the last visit being 12 (+/- 1.5) months from the day of surgery.
Arm/Group | Control | EVD Survivors
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/22
Other Adverse Events (participants affected / at risk) | 0/8 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=8) | EVD Survivors (N=22)
Subluxed intraocular lens (Eye disorders) | 1 (1) | 1 (1) — Subluxed intraocular lens with secondary anterior chambers lens placement at lens epithelial cell
Surgery on the fellow eye (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) — Inferior rhegmatogenous retinal detachment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03309020/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03309020/ICF_001.pdf